CLINICAL TRIAL: NCT04987151
Title: Comparison of Three Different Exercise Training Modalities (Aerobic, Strength, and Mixed) in Patients With Schizophrenia: Study Protocol for a Multi-centre Randomised Wait-list Controlled Trial
Brief Title: The Effects of Different Modalities of Exercise in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Laura García Garcés, Head of Nursing and Physiotherapy, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY UCH-CEU
Record Dates: First submitted 2021-07-19; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Strength training (Experimental): Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to strength training exercise involving the major muscle groups.
  Interventions: Other: Experimental-Strength training
- Aerobic training (Experimental): Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to brisk walking,
  Interventions: Other: Experimental-Aerobic training
- Strength/Aerobic training (Experimental): Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching), 15 minutes are allocated to brisk walking and 25 minutes are allocated to strength training involving the major muscle groups
  Interventions: Other: Experimental-Strength/Aerobic training
- Control Group (No Intervention): All the patients in the wait-list control group will receive one of the three trainings immediately after the intervention.

INTERVENTIONS:
Other: Experimental-Strength training — Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to strength training exercise involving the major muscle groups
  Arms: Strength training
Other: Experimental-Aerobic training — Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching) and 40 minutes are allocated to brisk walking.
  Arms: Aerobic training
Other: Experimental-Strength/Aerobic training — Each session lass 60 minutes, during which time 20 minutes are allocated for warming up and cooling down (stretching), 15 minutes are allocated to brisk walking and 25 minutes are allocated to strength training involving the major muscle groups.
  Arms: Strength/Aerobic training

SUMMARY:
Introduction: Numerous studies support the practice of different physical exercise modalities as an effective treatment to address the different problems associated with schizophrenia, reporting that they result in significant improvements in patient symptoms and quality of life. Given the lack of studies comparing different types of training in controlled environments, the aim of this proposed study will be to compare the effects of three physical exercise programs (strength, aerobic, and mixed) on the symptoms, body composition, level of physical activity, and health-related quality of life of patients with schizophrenia.

Ethics and dissemination: This study was approved by the ethics committees for Biomedical Research at the CEU Cardenal Herrera University of Valencia in Spain (reference number: CEI18/215). Participants will be fully informed of the purpose and procedures of the study, and written informed consent will be obtained from every participant. The results from this study will be published in peer-reviewed journals and presented in scientific conferences.

DETAILED DESCRIPTION:
The aim of this proposed study will be to compare the effects of three physical exercise programs (strength, aerobic, and mixed) on the symptoms, body composition, level of physical activity, and health-related quality of life of patients with schizophrenia.

A multicentre, single-blinded (evaluator), randomised, wait-list controlled (ratio 2:2:2:1) trial will be conducted with 105 patients recruited from different psychosocial care centres. The participants will be randomised into three 16-week training groups comprising 48 sessions lasting one hour each, or to the wait-list control group. The training groups will complete aerobic, strength, or mixed (aerobic + strength) training. The participants will be assessed before, immediately after, and 6 months after the end of the intervention. All the patients in the wait-list control group (n = 15) will receive one of the three trainings immediately after the intervention. The study variables will include positive symptomatology, negative symptomatology, and general symptomology (using the Positive and Negative Syndrome Scale) as the primary outcome; as secondary outcome: body composition (by assessing body mass index, body fat mass and waist circumference), physical activity levels (International Physical Activity Questionnaire-Short Form), and quality of life (abbreviated World Health Organization Quality of Life questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia
* Age between 18-65 years

Exclusion Criteria:

* Patients with other mental diseases
* Patients with mental disabilities
* Patients who present motor or behavioral pathologies that prevent the realization of the exercise training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 16 weeks
  Symptoms of schizophrenia are measured according to the subscale scores and total score on the PANSS which consists of 30 items scored from 1 (Absent) to 7 (Extreme). Scores range from 30 to 210, with higher scores indicating more symptoms

SECONDARY OUTCOMES:
World Health Organization Quality of Life-Short version (WHOQOL-BREF) | 16 weeks
  The WHOQOL-BREF contains 24 questions covering 4 domains plus two questions related to overall quality of life and satisfaction with health. Highes scores represent higher quality of life.
Body Mass Index (BMI) | 16 weeks
  The BMI is defined as the body mass divided by the square of the body height.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU-Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be available to other researchers.
Supporting Information: Study Protocol
Time Frame: Inmediately following publication.

REFERENCES:
- [Derived] Garcia-Garces L, Lacamara Cano S, Cebolla Melia Y, Sanchez-Lopez MI, Marques Azcona D, Lison JF, Peyro-Gregori L. Comparison of three different exercise training modalities (aerobic, strength and mixed) in patients with schizophrenia: study protocol for a multicentre randomised wait-list controlled trial. BMJ Open. 2021 Sep 17;11(9):e046216. doi: 10.1136/bmjopen-2020-046216. PMID 34535474